CLINICAL TRIAL: NCT06397456
Title: Intensive Patient Referral and Education Program Prior to Renal Replacement Therapy
Acronym: iPREP-RRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB20-1663; R01DK124597 (NIH)
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: Hospitalized Patients; African American; Motivational Interviewing
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — Blood Pressure Monitors; Self-Management

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The care provider will not be involved in the enrollment or assessment process. The outcomes assessor will analyze the outcomes without knowledge of allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Intervention (iPREP RRT) (Experimental): The intervention is administered by a patient educator (PE), a culturally concordant health educator. S/he will review the CKD and RRT education materials on a tablet device with the participant, answer any questions they have, and using motivational interviewing techniques get a commitment for future action. The participant and the patient educator will work together to decide on potential CKD self-management and RRT options and/or next steps. The PE will teach the participant how to use the home blood pressure monitor and will leave it with the participant.
  The patient educator will check in with the participant through text messages and follow-up phone calls.
  Interventions: Behavioral: In-Person Patient Education; Behavioral: Commitment to Change; Behavioral: Blood pressure monitoring; Behavioral: Text-based reinforcement for CKD self-management; Behavioral: Community-based education session, reinforcement for self-management
- Enhanced Usual Care (Placebo Comparator): The enhanced usual care is administered by a patient educator (PE), a culturally concordant health educator. The PE will drop off written general health education materials.
  The patient educator will check in with the participant through text messages.
  Interventions: Behavioral: Written Patient Education; Behavioral: Text-based reinforcement for general health self-management

INTERVENTIONS:
Behavioral: In-Person Patient Education — In-person patient education about CKD, CKD risk factor management and renal replacement therapy options.
  Arms: Intensive Intervention (iPREP RRT)
Behavioral: Commitment to Change — Motivational interviewing to assist participants in committing to change in CKD management or RRT selection.
  Arms: Intensive Intervention (iPREP RRT)
Behavioral: Blood pressure monitoring — Participants will learn how to check their blood pressure and will receive a blood pressure cuff for home.
  Arms: Intensive Intervention (iPREP RRT)
Behavioral: Written Patient Education — Written patient education booklet about general health care management including taking medications, having a primary care doctor, weight management and exercise.
  Arms: Enhanced Usual Care
Behavioral: Text-based reinforcement for CKD self-management — Patient educator will use text messages based on social cognitive theory to remind participants about and reinforce goals set around CKD self-management, blood pressure control and RRT selection
  Arms: Intensive Intervention (iPREP RRT)
Behavioral: Community-based education session, reinforcement for self-management — Patient educator will use provide a "booster" session based on social cognitive theory to remind participants about and reinforce goals set around CKD self-management, blood pressure control and RRT selection
  Arms: Intensive Intervention (iPREP RRT)
Behavioral: Text-based reinforcement for general health self-management — Patient educator will use text messages to send general health management messages
  Arms: Enhanced Usual Care

SUMMARY:
Intensive Patient Referral and Education Program prior to Renal Replacement Therapy (iPREP-RRT) is a 12-week intervention that identifies hospitalized African Americans with advanced chronic kidney disease (CKD) and provides them with hospital- and community-based education, navigation and self-management support. Participants will be randomized to the iPREP-RRT intervention versus enhanced usual care.

DETAILED DESCRIPTION:
The Intensive Patient Referral and Education Program prior to Renal Replacement Therapy (iPREP-RRT) will determine the efficacy of the hospital-based patient intervention (HPI) in improving patient knowledge, self-efficacy, and intent for chronic kidney disease (CKD) self-management and renal replacement therapy (RRT) planning; and 2) determine the efficacy of the community-based patient intervention (CPI) during a 12 week outpatient follow-up program that combines outpatient follow-up with multiple modes of communication (in-person session, phone calls and personalized text messaging) and navigation in increasing participants' initiation and maintenance of CKD self-management and RRT planning, compared to enhanced usual care (attention controls).

The goal is to improve knowledge and outcomes for African American patients with advanced CKD through the iPREP-RRT. To accomplish this goal, investigators will 1) determine the efficacy of the hospital-based patient intervention (HPI) in improving participant knowledge, self-efficacy, and intent for CKD self-management and RRT planning; and 2) determine the efficacy of the community-based patient intervention (CPI) during a 12 week outpatient program that combines outpatient follow-up with multiple modes of communication (in-person session, phone calls and personalized text messaging) and navigation in increasing initiation and maintenance of CKD self-management and RRT planning, compared to enhanced usual care. To that end, investigators will conduct a one-site randomized controlled trial, where participants will be randomized in a 1:1 ratio into either the intervention (iPREP-RRT) or control groups (enhanced usual care). The randomization will be stratified by baseline blood pressure (controlled or uncontrolled). Participants will receive 2 in-person education sessions (during hospitalization and week 12), phone sessions at weeks 4 and 8, and weekly personalized text message contact. The duration of the intervention will be 12 weeks, and participants and controls will be assessed pre-intervention, immediately post-hospital based intervention, at 4 ,8 and 12 weeks during community-based intervention and 4 weeks post-intervention (16 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 and under 70
* Admitted to the University of Chicago inpatient general medicine service
* Likely hospital stay greater than 48 hours
* Diagnosis of advanced CKD (Stage 3B or above, as determine by problem list, ICD- 10 codes or eGFR<45 during admission and from previous medical encounters)
* Self-identify as Black or African American

Exclusion Criteria:

* Non-English speaking
* Unable to communicate due to current medical status
* Unable to consent due to mental status
* Expected hospital stay less than 24 hour
* Current admission in ICU

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Kidney Disease Knowledge Questionnaire (KIKS) | Baseline, 1 day Post Brief Intervention, Week 4, Week 12, Week 16
  The Kidney Disease Knowledge Questionnaire (KIKS) is a validated instrument that assesses CKD knowledge. Scores range from 0 (no knowledge)-28 (full knowledge). Change =Post intervention-Baseline scores, and Follow-up (Week 4, Week 12, Week 16)-Baseline
ESRD Knowledge | Baseline, 1 day Post Brief Intervention, Week 4, Week 12, Week 16
  The Kidney Failure Treatment Knowledge is an investigator developed tool that assesses knowledge of 6 ESKD treatment options using a Likert scale (0=no knowledge and 4=a great deal of knowledge). Possible scores range from 0-24. Change =Post intervention-Baseline scores, and Follow-up (Week 4, Week 12, Week 16)-Baseline
Blood Pressure Knowledge | Baseline, 1 day Post Brief Intervention, Week 4, Week 12, Week 16
  Blood Pressure Knowledge Scale (BPKS, revised) is an 11-item scale; a summed score is computed. Scores range from 7 to 77 and higher scores indicate greater knowledge. Change =Post intervention-Baseline scores, and Follow-up (Week 4, Week 12, Week 16)-Baseline
CKD Self-Management | Baseline, Week 8, Week 12, Week 16
  The CKD Self-Management Knowledge Toolkit (CKD-SMKT) is a validated 10 item survey to assess participants CKD self-management behaviors. The survey consists of 2 true /false questions for each of the 10 self-care domains and can be scored from 0 (no self-care) to 20 (full self-care). Change is Follow-up Score (Week 8, Week 12, Week 16)-Baseline

SECONDARY OUTCOMES:
CKD Self-Efficacy | Baseline, 1 day Post Brief Intervention, Week 4, Week 8, Week 12, Week 16
  CKD Self-Efficacy Scale (CKD-SE), 25-item CKD-SE instrument can be used for the early identification of patients with low self-efficacy. The scale is from 0 to 10 points, and a larger number indicates a higher level of confidence regarding the management activity. The total score on the scale ranges between 25 and 250. The total score can be classified into three categories: low self-efficacy (score less than 30), moderate (scores between 30 to 70), and high self-efficacy (score more than 70). Change is Follow-up Score (Week 8, Week 12, Week 16)-Baseline
CKD Health Intent | Baseline, 1 day Post-Brief Intervention, Week 4
  The Health Intent Survey is an investigator-developed tool to measure participants stated intent to make healthy lifestyle changes. There are 12 questions each scored on a 5 point scale from 1=extremely unlikely to 5=extremely likely (60 total possible points with higher scores better). Change=Follow-up (1 day post-intervention, Wk4, wk 8, wk 12, wk16) - baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Will share de-identified, aggregate data with other researchers. Additional sharing not permitted by current IRB permission.